CLINICAL TRIAL: NCT05561387
Title: A Phase III Randomized Trial for Newly Diagnosed Multiple Myeloma (NDMM) Patients Considered Frail or in a Subset of "Intermediate Fit" Comparing Upfront Three-Drug Induction Regimens Followed by Double or Single-Agent Maintenance
Brief Title: Comparing Combinations of Drugs to Treat Newly Diagnosed Multiple Myeloma (NDMM) When a Stem Cell Transplant is Not a Medically Suitable Treatment
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S2209; NCI-2022-05722 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S2209 (Other: SWOG); S2209 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2022-09-27; First posted 2022-09-30 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; daratumumab; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Arm I (VRd-Lite) (Active Comparator): INDUCTION CYCLES 1-9: Patients receive bortezomib SC on days 1, 8, 15, and 22 of each cycle, lenalidomide PO on days 1-21 of each cycle, and dexamethasone PO on days 1, 8, 15, and 22 of each cycle. Treatment repeats every 28 days for up to 9 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE CYCLES 10+: Patients receive lenalidomide PO on days 1-21 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bortezomib; Drug: Dexamethasone; Drug: Lenalidomide; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (DRd-R) (Experimental): INDUCTION CYCLES 1-9: Patients receive daratumumab and hyaluronidase-fihj SC on days 1, 8, 15, and 22 of cycles 1-2, days 1 and 15 of cycles 3-6, and day 1 of cycles 7-9, lenalidomide PO on days 1-21 of each cycle, and dexamethasone PO on days 1, 8, 15, and 22 of each cycle. Treatment repeats every 28 days for up to 9 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE CYCLES 10+: Patients receive lenalidomide PO on days 1-21 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Daratumumab and Hyaluronidase-fihj; Drug: Dexamethasone; Drug: Lenalidomide; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm III (DRd-DR): (Experimental): INDUCTION CYCLES 1-9: Patients receive daratumumab and hyaluronidase-fihj SC on days 1, 8, 15, and 22 of cycles 1-2, days 1 and 15 of cycles 3-6, and day 1 of cycles 7-9, lenalidomide PO on days 1-21 of each cycle, and dexamethasone PO on days 1, 8, 15, and 22 of each cycle. Treatment repeats every 28 days for up to 9 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE CYCLES 10+: Patients receive daratumumab and hyaluronidase-fihj SC on day 1 of each cycle and lenalidomide PO on days 1-21 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Daratumumab and Hyaluronidase-fihj; Drug: Dexamethasone; Drug: Lenalidomide; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Bortezomib — Given SC
  Other Names: [(1R)-3-Methyl-1-[[(2S)-1-oxo-3-phenyl-2-[(pyrazinylcarbonyl)amino]propyl]amino]butyl]boronic Acid; LDP 341; MLN341; PS-341; PS341; Velcade
  Arms: Arm I (VRd-Lite)
Drug: Daratumumab and Hyaluronidase-fihj — Given SC
  Other Names: DARA Co-formulated with rHuPH20; DARA/rHuPH20; Daratumumab + rHuPH20; Daratumumab with rHuPH20; Daratumumab-rHuPH20; Daratumumab/Hyaluronidase-fihj; Daratumumab/rHuPH20 Co-formulation; Darzalex Faspro; Darzalex/rHuPH20; HuMax-CD38-rHuPH20; Recombinant Human Hyaluronidase Mixed with Daratumumab
  Arms: Arm II (DRd-R); Arm III (DRd-DR):
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase III trial compares three-drug induction regimens followed by double-or single-drug maintenance therapy for the treatment of newly diagnosed multiple myeloma in patients who are not receiving a stem cell transplant and are considered frail or intermediate-fit based on age, comorbidities, and functional status. Treatment for multiple myeloma includes initial treatment (induction) which is the first treatment a patient receives for cancer followed by ongoing treatment (maintenance) which is given after initial treatment to help keep the cancer from coming back. There are three combinations of four different drugs being studied. Bortezomib is one of the drugs that may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Lenalidomide works by helping bone marrow to produce normal blood cells and killing cancer cells. Anti-inflammatory drugs, such as dexamethasone, lower the body's immune response and are used with other drugs in the treatment of some types of cancer. Daratumumab and hyaluronidase-fihj is a monoclonal antibody that may interfere with the ability of cancer cells to grow and spread. Patients receive 1 of 3 combinations of these drugs for treatment to determine which combination of study drugs works better to shrink and control multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare progression-free survival (PFS) in frail or selected intermediate fit newly diagnosed multiple myeloma (NDMM) participants treated with bortezomib with lenalidomide and dexamethasone at reduced dosing (VRd-Lite) induction followed by lenalidomide maintenance (Arm 1) versus daratumumab and hyaluronidase-fihj with lenalidomide and dexamethasone (DRd) induction followed by lenalidomide maintenance (Arm 2).

II. To compare overall survival (OS) in frail or selected intermediate fit NDMM participants treated with VRd-Lite induction followed by lenalidomide maintenance (Arm 1) versus DRd induction followed by lenalidomide and daratumumab and hyaluronidase-fihj maintenance (Arm 3).

SECONDARY OBJECTIVES:

I. To compare PFS in Arm 1 versus Arm 3 II. To compare OS in Arm 1 versus Arm 2. III. To compare PFS in Arm 2 versus 3. IV. To compare the overall response rate (ORR) of Arm 1 against the ORR of Arm 2 and Arm 3.

V. To compare the safety of Arm 1 with the safety of Arm 2 and Arm 3. VI. To explore veinous thrombo-embolism (VTE) incidence in participants receiving lenalidomide during induction across the three study arms.

VII. To describe median time to response (complete response [CR] or better per International Myeloma Working Group [IMWG] criteria, very good partial response [VGPR] or better per IMWG criteria, partial response [PR] or better per IMWG criteria) on the three study arms.

PRIMARY QUALITY OF LIFE (QOL) OBJECTIVE:

I. To compare patient-reported global health status between treatment arms (Arm 1 versus the combination of Arms 2 and 3) at 9 months after randomization (end of induction therapy) using the European Organization for Research and Treatment of Cancer (EORTC) Core Quality of Life Questionnaire (QLQ-C30).

SECONDARY QOL OBJECTIVE:

II. To compare longitudinal changes in global health status between treatment arms (Arm 1 versus the combination of Arms 2 and 3) from baseline to 9 months after randomization (end of induction therapy).

PATIENT REPORTED OUTCOMES-COMMON TERMINOLOGY CRITERIA FOR ADVERSE EVENTS (PRO-CTCAE) OBJECTIVE:

I. To compare selected patient-reported outcome symptoms using PRO-CTCAE items among the 3 study arms.

ADDITIONAL OBJECTIVES:

I. To compare the rate of minimal residual disease (MRD) by clonoSEQ after 9 cycles of induction in Arm 1 versus Arm 2 and Arm 3, respectively.

II. To compare the rate of MRD conversion after 1 year of maintenance in participants who were MRD positive after induction in Arm 1 versus Arm 2 and Arm 3, respectively.

III. To compare the rate of sustained MRD negativity at time points of post-induction, post-1 year maintenance in Arm 1 versus Arm 2 and Arm 3, respectively.

BANKING OBJECTIVES:

I. To bank specimens for future correlative studies.

OUTLINE: Patients are randomized to 1 of 3 arms.

ARM I (VRd-Lite):

INDUCTION CYCLES 1-9: Patients receive bortezomib subcutaneously (SC) on days 1, 8, 15, and 22 of each cycle, lenalidomide orally (PO) on days 1-21 of each cycle, and dexamethasone PO on days 1, 8, 15, and 22 of each cycle. Treatment repeats every 28 days for up to 9 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE CYCLES 10+: Patients receive lenalidomide PO on days 1-21 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM II (DRd-R):

INDUCTION CYCLES 1-9: Patients receive daratumumab and hyaluronidase-fihj SC on days 1, 8, 15, and 22 of cycles 1-2, days 1 and 15 of cycles 3-6, and day 1 of cycles 7-9, lenalidomide PO on days 1-21 of each cycle, and dexamethasone PO on days 1, 8, 15, and 22 of each cycle. Treatment repeats every 28 days for up to 9 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE CYCLES 10+: Patients receive lenalidomide PO on days 1-21 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM III (DRd-DR):

INDUCTION CYCLES 1-9: Patients receive daratumumab and hyaluronidase-fihj SC on days 1, 8, 15, and 22 of cycles 1-2, days 1 and 15 of cycles 3-6, and day 1 of cycles 7-9, lenalidomide PO on days 1-21 of each cycle, and dexamethasone PO on days 1, 8, 15, and 22 of each cycle. Treatment repeats every 28 days for up to 9 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE CYCLES 10+: Patients receive daratumumab and hyaluronidase-fihj SC on day 1 of each cycle and lenalidomide PO on days 1-21 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year, every 6 months for 2 years, and then annually for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have documented multiple myeloma satisfying standard International Myeloma Working Group (IMWG) diagnostic criteria within 28 days prior to registration
* Participants must have measurable disease within 28 days prior to registration as defined by any of the following:

  * Immunoglobulin (Ig) G myeloma (serum monoclonal paraprotein [M-protein] level >= 0.5 gram/deciliter [g/dL] or urine M-protein level >= 200 milligram[mg]/24 hours[hrs]); OR
  * IgA, IgM, IgD, or IgE multiple myeloma (serum M-protein level >= 0.2 g/dL or urine M-protein level >= 200 mg/24 hrs); OR
  * Light chain multiple myeloma (serum immunoglobulin free light chain >= 10 mg/dL and abnormal serum immunoglobulin kappa lambda free light chain ratio)
* All disease must be assessed and documented on the baseline/pre-registration tumor assessment form
* Participants must have a calculated myeloma frailty index (Myeloma Frailty Score Calculator; http://www.myelomafrailtyscorecalculator.net/) categorized as frail or intermediate fit (regardless of age) within 28 days prior to registration
* For Participants Meeting "Frail" Status:

  * Participants with any degree of kidney dysfunction are allowed; however, participants on dialysis are not eligible
* For Participants Meeting "Frail" Status:

  * Hemoglobin >= 7 g/dL (must be performed within 28 days prior to registration)

    * Note: growth factor and transfusion utilization are allowed if cytopenias are considered secondary to bone marrow involvement from MM)
* For Participants Meeting "Frail" Status:

  * Platelets >= 50 x 10^9/L (must be performed within 28 days prior to registration)

    * Note: growth factor and transfusion utilization are allowed if cytopenias are considered secondary to bone marrow involvement from MM)
* For Participants Meeting "Frail" Status:

  * Absolute neutrophil count (ANC) >= 0.75 x10^9/L (must be performed within 28 days prior to registration)

    * Note: growth factor and transfusion utilization are allowed if cytopenias are considered secondary to bone marrow involvement from MM)
* For Participants Meeting "Intermediate Fit" Status, one or more of the following criteria must be present:

  * Kidney dysfunction showing calculated creatinine clearance (CrCl) <30 ml/min.

    * Actual lab serum creatinine value with a minimum of 0.7 mg/dL.
  * Participants must have bone marrow function assessed and meet the below criteria ranges:

    * Hemoglobin between 7-8 g/dL, OR
    * Platelets between 50-75 x10^9/L, OR
    * ANC between 0.75-1 x10^9/L

      * Note: growth factor and transfusion utilization are allowed as long as cytopenias are considered secondary to bone marrow involvement from MM)
  * Revised International Staging System (R-ISS) stage III disease
  * Note: All labs must be performed within 28 days prior to registration
* Participants must have a complete medical history and physical exam within 28 days prior to registration
* Participants must have whole body imaging within 60 days prior to registration. The recommended method of imaging is a positron emission tomography/computed tomography (PET/CT); a low-dose whole body CT scan or whole-body magnetic resonance imaging (MRI) or skeletal survey should be done only if a PET/CT scan cannot be done or is non-feasible. This must be documented in the comments section of the Onstudy form.
* Total bilirubin =< 2 times institutional upper limit of normal (ULN) unless history of Gilbert's disease. Participants with history of Gilbert's disease must have total bilirubin =< 5 x institutional ULN (within 28 days prior to registration)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 3 × institutional ULN (within 28 days prior to registration)
* Participants must have adequate cardiac function, as assessed by the treating physician within 14 days prior to registration. Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, must have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification and must not be assessed as class 3 or 4
* Participants with known diabetes must show evidence of controlled disease within 14 days prior to registration. Uncontrolled diabetes is defined as: A glycosylated hemoglobin (Hg)A1C > 7
* Participants with known human immunodeficiency virus (HIV)-infection must be receiving anti-retroviral therapy and have an undetectable viral load test on the most recent test result obtained, within 6 months prior to registration
* All participants with evidence of chronic hepatitis B virus (HBV) infection must have undetectable HBV viral load on suppressive therapy within 28 days prior to registration
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. For participants with HCV infection who are currently on treatment, participant must have an undetectable HCV viral load within 28 days prior to registration
* Participants must have an Eastern Cooperative Oncology Group (ECOG)/Zubrod performance status score of 0-2 (Note: Participants with ECOG/Zubrod performance score [PS] 3, especially where the deterioration of PS is considered secondary to the MM diagnosis, will be allowed)
* Participants must be offered the opportunity to participate in specimen banking. With participant consent, specimens must be collected and submitted via the Southwest Oncology Group (SWOG) specimen tracking system
* Participants who are able to complete the patient-reported outcomes measures in English or Spanish must agree to participate in the PRO portion of the study
* Participants must be informed of the investigational nature of this study and must sign and give informed consent in accordance with institutional and federal guidelines. For participants with impaired decision-making capabilities, legally authorized representatives may sign and give informed consent on behalf of study participants in accordance with applicable federal, local, and Central Institutional Review Board (CIRB) regulations

Exclusion Criteria:

* Participants must not have received any prior systemic therapy for multiple myeloma with the exception of any one or more of the following:

  * An emergency use of a short course of corticosteroids (equivalent of dexamethasone 160 mg) any time before registration, or
  * Up to one complete cycle of a non-daratumumab and hyaluronidase-fihj containing anti-myeloma regimen (1 cycle = 21 or 28 days depending on the regimen being used), or
  * Localized palliative radiation therapy for multiple myeloma, as long as the radiation therapy is completed at least 3 days prior to starting the systemic treatment as per the study protocol.
* Participants must not have evidence of grade 4 peripheral neuropathy prior to study registration
* Participants must not have uncontrolled blood pressure within 14 days prior to registration. Uncontrolled blood pressure: systolic blood pressure (SBP) > 140 mmHg or diastolic blood pressure (DBP) > 90 mmHg. Participants are permitted to be receiving multiple anti-hypertensive medications (unless otherwise indicated in the study). All blood pressure measurements within the 14 days prior to registration must be SBP =< 140 and DBP =< 90. A participant with a single blood pressure elevation who upon rechecking has a normal blood pressure will remain eligible at the discretion of the registering investigator.
* Participants must not have a prior or concurrent malignancy whose natural history or treatment (in the opinion of the treating physician) has the potential to interfere with the safety or efficacy assessment of the investigational regimen.
* Participants must not be pregnant or nursing. Individuals who are of reproductive potential must have agreed to use an effective contraceptive method with details provided as a part of the consent process. A person who has had menses at any time in the preceding 24 consecutive months or who has semen likely to contain sperm is considered to be of "reproductive potential." In addition to routine contraceptive methods, "effective contraception" also includes refraining from sexual activity that might result in pregnancy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) including hysterectomy, bilateral oophorectomy, bilateral tubal ligation/occlusion, and vasectomy with testing showing no sperm in the semen.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 510 (Estimated)
Dates: Start 2023-10-12 (Actual); Primary Completion 2031-05-30 (Estimated); Study Completion 2031-05-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) of Arm 1 versus (vs.) Arm 2 | From date of randomization to date of first documentation of progression or symptomatic deterioration, or death due to any cause, or assessed up to 10 years
  Analysis of each of the dual primary endpoints will be performed using a stratified log-rank test for comparison between arms. The analyses will be stratified according to frailty score (frail vs. intermediate fit), presence of one or more high-risk abnormalities by fluorescence in situ hybridization (iFISH) (yes vs. no), and prior therapy (yes vs. no). All eligible participants will be considered in analyses of the dual primary endpoints, according to their assigned arm at randomization.
Overall survival (OS) of Arm 1 vs. Arm 3 | From date of randomization to date of death due to any cause, or assessed up to 10 years
  Analysis of each of the dual primary endpoints will be performed using a stratified log-rank test for comparison between arms. The analyses will be stratified according to frailty score (frail vs. intermediate fit), presence of one or more high-risk abnormalities by iFISH (yes vs. no), and prior therapy (yes vs. no). All eligible participants will be considered in analyses of the dual primary endpoints, according to their assigned arm at randomization.

SECONDARY OUTCOMES:
PFS | From date of randomization to date of first documentation of progression or symptomatic deterioration, or death due to any cause, or assessed up to 10 years
  Analysis of PFS and OS endpoints will be performed using a stratified log-rank test for comparison between arms, with stratification according to frailty score (frail vs. intermediate fit) presence of one or more high-risk abnormalities by iFISH (yes vs. no) and prior therapy (yes vs. no).
OS | From date of randomization to date of death due to any cause, or assessed up to 10 years
  Analysis of PFS and OS endpoints will be performed using a stratified log-rank test for comparison between arms, with stratification according to frailty score (frail vs. intermediate fit) presence of one or more high-risk abnormalities by iFISH (yes vs. no) and prior therapy (yes vs. no).
Overall response rate (ORR) | Up to 10 years
  ORR is defined as the percentage of participants achieving a best response of partial response (PR) or better while on study. ORR will be reported with a binomial confidence interval. Time to response will be analyzed using the cumulative incidence competing risks method.
Time to complete response (CR) | The time from the date of registration to the date of the first documented incidence of a response of CR or better, assessed up to 10 years
  All eligible participants will be considered in analyses of the secondary endpoints, according to their assigned arm at randomization, and with participants who go off-study prior to response assessment considered as non-responders for the analysis of response rate and as censored at the time of removal from study for the analysis of time to response. Time to response will be analyzed using the cumulative incidence competing risks method.
Time to very good partial response (VGFR) | The time from the date of registration to the date of the first documented incidence of a response of VGPR or better, assessed up to 10 years
  All eligible participants will be considered in analyses of the secondary endpoints, according to their assigned arm at randomization, and with participants who go off-study prior to response assessment considered as non-responders for the analysis of response rate and as censored at the time of removal from study for the analysis of time to response. Time to response will be analyzed using the cumulative incidence competing risks method.
Time to PR | The time from the date of registration to the date of the first documented incidence of a response of PR or better, assessed up to 10 years
  All eligible participants will be considered in analyses of the secondary endpoints, according to their assigned arm at randomization, and with participants who go off-study prior to response assessment considered as non-responders for the analysis of response rate and as censored at the time of removal from study for the analysis of time to response. Time to response will be analyzed using the cumulative incidence competing risks method.
Minimal residual disease (MRD) | At 9 months of induction therapy and 1 year of maintenance therapy
  The rate of MRD negativity will be calculated at each timepoint as the number of patients who are MRD negative divided by the number of patients who were eligible, analyzable and assessable for clinical response assessment at that timepoint. Rates of MRD negativity will be compared using a two-arm binomial test.
Patient report out comes (PRO) quality-of-life (QOL) | At baseline and months 1, 3, 9, and 18 after randomization
  We will use the European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 (version 3). This instrument includes questions broadly applicable to all cancer patients, assessing 5 functional domains (physical, role, cognitive, emotional, social) and 8 symptoms (fatigue, pain, nausea/vomiting, dyspnea, loss of appetite, insomnia, constipation, diarrhea), together with financial problems and global quality of life.
Patient-reported toxicity (PRO-Common Terminology Criteria for Adverse Events [CTCAE]) | At baseline, at each treatment cycle up to month 18 from randomization, and at discontinuation of treatment
  PRO-CTCAE is intended to enhance the quality of adverse event data reporting in clinical trials, provide data that complements and extends the information provided by clinician reporting using CTCAE, represent the patient perspective of the experience of symptomatic adverse events (AEs), and improve detection of potentially serious adverse events. Descriptive statistics will be used to summarize selected PRO-CTCAEs tabulated at each cycle overall and by arm. We will examine the extent to which PRO-CTCAEs with provider reported AEs are correlated and evaluate differences in incidence and worst severity.

CONTACTS AND LOCATIONS:
Overall Officials: Sikander Ailawadhi, Principal Investigator — SWOG Cancer Research Network
Locations (397):
- United States (397):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CARTI Cancer Center, Little Rock, Arkansas
  - John L McClellan Memorial Veterans Hospital, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Marshall Cancer Center, Cameron Park, California
  - Mercy Cancer Center - Carmichael, Carmichael, California
  - Mercy San Juan Medical Center, Carmichael, California
  - Mercy Cancer Center - Elk Grove, Elk Grove, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Mercy UC Davis Cancer Center, Merced, California
  - Providence Queen of The Valley, Napa, California
  - Mercy Cancer Center - Rocklin, Rocklin, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Providence Medical Foundation - Santa Rosa, Santa Rosa, California
  - Providence Santa Rosa Memorial Hospital, Santa Rosa, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Woodland Memorial Hospital, Woodland, California
  - Rocky Mountain Regional VA Medical Center, Aurora, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Saint Francis Cancer Center, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center at Glastonbury, Glastonbury, Connecticut
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital Care Center at Long Ridge, Stamford, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Saint Anthony's Health, Alton, Illinois
  - Rush - Copley Medical Center, Aurora, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Loyola Center for Health at Burr Ridge, Burr Ridge, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Saint Mary's Hospital, Centralia, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Edward Hines Jr VA Hospital, Hines, Illinois
  - Loyola Medicine Homer Glen, Homer Glen, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Marjorie Weinberg Cancer Center at Loyola-Gottlieb, Melrose Park, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - IU Health North Hospital, Carmel, Indiana
  - Northwest Cancer Center - Main Campus, Crown Point, Indiana
  - Northwest Oncology LLC, Dyer, Indiana
  - Northwest Cancer Center - Hobart, Hobart, Indiana
  - Saint Mary Medical Center, Hobart, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Saint Catherine Hospital, Indianapolis, Indiana
  - The Community Hospital, Munster, Indiana
  - Women's Diagnostic Center - Munster, Munster, Indiana
  - Reid Health, Richmond, Indiana
  - Northwest Cancer Center - Valparaiso, Valparaiso, Indiana
  - Mission Cancer and Blood - Ankeny, Ankeny, Iowa
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Mission Cancer and Blood - Laurel, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Hospital, Lexington, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Saint Joseph Mount Sterling, Mount Sterling, Kentucky
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Great Lakes Cancer Management Specialists-Doctors Park, East China Township, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Academic Hematology Oncology Specialists, Grosse Pointe Woods, Michigan
  - Great Lakes Cancer Management Specialists-Van Elslander Cancer Center, Grosse Pointe Woods, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Ascension Borgess Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Medical Campus, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - 21st Century Oncology-Pontiac, Pontiac, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Ascension Saint Joseph Hospital, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Professional Building, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Michigan Breast Specialists-Warren, Warren, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Riverwood Healthcare Center, Aitkin, Minnesota
  - Essentia Health - Baxter Clinic, Baxter, Minnesota
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Essentia Health - Ely Clinic, Ely, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Essentia Health - International Falls Clinic, International Falls, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - Essentia Health - Moose Lake Clinic, Moose Lake, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Sanford Cancer Center Worthington, Worthington, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Lake Regional Hospital, Osage Beach, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Exeter Hospital, Exeter, New Hampshire
  - Lovelace Medical Center-Saint Joseph Square, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Presbyterian Rust Medical Center/Jorgensen Cancer Center, Rio Rancho, New Mexico
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford South University Medical Center, Fargo, North Dakota
  - Southpointe-Sanford Medical Center Fargo, Fargo, North Dakota
  - Sanford Medical Center Fargo, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Essentia Health - Jamestown Clinic, Jamestown, North Dakota
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Saint Elizabeth Boardman Hospital, Boardman, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Dayton Physician LLC-Miami Valley Hospital North, Dayton, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Saint Joseph Warren Hospital, Warren, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Rogue Valley Medical Center, Medford, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Smilow Cancer Hospital Care Center - Westerly, Westerly, Rhode Island
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Avera Cancer Institute-Aberdeen, Aberdeen, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Avera Cancer Institute at Yankton, Yankton, South Dakota
  - MD Anderson in The Woodlands, Conroe, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Michael E DeBakey VA Medical Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - MD Anderson League City, League City, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - Sovah Health Martinsville, Martinsville, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Essentia Health-Hayward Clinic, Hayward, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Clinic - Ladysmith Center, Ladysmith, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aspirus Medford Hospital, Medford, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Marshfield Medical Center - Neillsville, Neillsville, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Ascension Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Essentia Health-Spooner Clinic, Spooner, Wisconsin
  - Ascension Saint Michael's Hospital, Stevens Point, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Essentia Health Saint Mary's Hospital - Superior, Superior, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin